CLINICAL TRIAL: NCT02909582
Title: Obesity: Cesarean Health by Incision Placement
Acronym: O-CHIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Rebekah McCurdy, Obstetrician/Maternal Fetal Medicine Fellow, Thomas Jefferson University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16D.541
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Maternal Morbidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pfannenstiel Incision (No Intervention): This curved incision is approximately 10-15 cm long and 2 cm above the pubic symphysis. If a pannus is present, the pannus should be retracted up (see diagram) to allow placement of the Pfannenstiel incision.
- Cohen Incision (Experimental): This is a straight transverse incision through the skin, 3 cm below the level of the anterior superior iliac spines (higher than the Pfannenstiel incision). Should a pannus exist, the pannus should be left in the physiologic location (not retracted) to allow placement of the incision.
  Interventions: Procedure: Cohen Incision

INTERVENTIONS:
Procedure: Cohen Incision — This is a straight transverse incision through the skin, 3 cm below the level of the anterior superior iliac spines (higher than the Pfannenstiel incision). Should a pannus exist, the pannus should be left in the physiologic location (not retracted) to allow placement of the incision.
  Arms: Cohen Incision

SUMMARY:
Hypothesis: A Pfannenstiel cesarean skin incision placed under the pannus (should a pannus exist) will have a higher maternal morbidity composite rate than a Cohen cesarean skin incision placed above the pannus (should a pannus exist).

DETAILED DESCRIPTION:
Introduction: Obesity affects approximately 1/3rd of all reproductive-aged women and is associated with increased maternal morbidity during and after cesarean section. The optimal surgical approach has not been well elucidated for obese individuals.

Materials and Methods: This is a randomized controlled trial comparing a Pfannenstiel incision placed below the pannus (should a pannus exist) with a Cohen incision placed above the pannus (should a pannus exist); allocation is 1:1 with stratification for pre-gestational diabetes and presence of pannus. The study will be assessed by intention-to-treat analysis looking composite maternal morbidity (wound complications within 6 weeks, endometritis, postpartum hemorrhage) as the primary outcome with secondary outcomes including wound complications, operative time, estimated blood loss, pain management, and patient and surgeon satisfaction. Significant confounders will be assessed and adjusted in the multiple regression analysis accordingly.

Results: The investigators propose the Cohen cesarean incision will result in statistically less maternal morbidity from cesarean section than the Pfannenstiel incision.

Comment: The benefits of a Cohen incision have been encouraged in non-obese pregnant women; the investigators propose that they be considered in obese women as well.

ELIGIBILITY:
Inclusion Criteria:

* BMI > or = 35 kg/m2 at time of presentation for delivery
* Speaks English

Exclusion Criteria:

* BMI < 35 kg/m2 at time of presentation or delivery
* Unable to consent (including language spoken other than English)
* Prior abdominal incisions or obstetric factors necessitating placement of incision in specified location, at the discretion of the attending surgeon
* Infection present (ie cellulitis) precluding incision placement at one of the randomization sites

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 284 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Composite Maternal Morbidity | 18 months
  To compare composite maternal morbidity (wound complications within 6 weeks including cellulitis, wound abscess, wound separation or dehiscence, hematoma, seroma formation, endometritis, postpartum hemorrhage), by placement type of transverse Cesarean skin incision in individuals with BMI >35 kg/m2.

SECONDARY OUTCOMES:
Composite maternal morbidity (as above) by stage of pannus | 18 months
Composite wound complication rates (cellulitis, wound abscess, wound separation or dehiscence, hematoma, seroma) | 18 months
Length in minutes of operative time from time of skin incision to time of delivery of the neonate | 18 months
Length in minutes of total operating time (from time of skin incision to the completion of closure of the skin incision) | 18 months
Patient satisfaction (via two questions, Likert scale) | 18 months
Severity of pain (via Likert scale) and amount of pain medications utilized in the first 48 hours post procedure | 18 months
Estimated blood loss (in milliliters) | 18 months
Incidence of low transverse uterine incisions (hysterotomy) with all other types of uterine incisions (vertical, high transverse, etc). | 18 months
Attending surgeon satisfaction (on 1-10 Likert scale) with feasibility of surgery by incision type | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hofmeyr JG, Novikova N, Mathai M, Shah A. Techniques for cesarean section. Am J Obstet Gynecol. 2009 Nov;201(5):431-44. doi: 10.1016/j.ajog.2009.03.018. PMID 19879392
- [Background] Chu SY, Kim SY, Schmid CH, Dietz PM, Callaghan WM, Lau J, Curtis KM. Maternal obesity and risk of cesarean delivery: a meta-analysis. Obes Rev. 2007 Sep;8(5):385-94. doi: 10.1111/j.1467-789X.2007.00397.x. PMID 17716296
- [Background] Ayres-de-Campos D. Obesity and the challenges of caesarean delivery: prevention and management of wound complications. Best Pract Res Clin Obstet Gynaecol. 2015 Apr;29(3):406-14. doi: 10.1016/j.bpobgyn.2014.08.009. Epub 2014 Oct 16. PMID 25457856
- [Background] Houston MC, Raynor BD. Postoperative morbidity in the morbidly obese parturient woman: supraumbilical and low transverse abdominal approaches. Am J Obstet Gynecol. 2000 May;182(5):1033-5. doi: 10.1067/mob.2000.105400. PMID 10819819
- [Background] Wall PD, Deucy EE, Glantz JC, Pressman EK. Vertical skin incisions and wound complications in the obese parturient. Obstet Gynecol. 2003 Nov;102(5 Pt 1):952-6. doi: 10.1016/s0029-7844(03)00861-5. PMID 14672469
- [Background] Alanis MC, Villers MS, Law TL, Steadman EM, Robinson CJ. Complications of cesarean delivery in the massively obese parturient. Am J Obstet Gynecol. 2010 Sep;203(3):271.e1-7. doi: 10.1016/j.ajog.2010.06.049. Epub 2010 Aug 3. PMID 20678746
- [Background] Marrs CC, Moussa HN, Sibai BM, Blackwell SC. REMOVED: The relationship between primary cesarean delivery skin incision type and wound complications in women with morbid obesity. Am J Obstet Gynecol. 2014 Apr;210(4):319. doi: 10.1016/j.ajog.2014.01.018. Epub 2014 Feb 20. PMID 24560557 (Retraction: PMID 28648694 Am J Obstet Gynecol. 2017 Jul;217(1):85)